CLINICAL TRIAL: NCT02675400
Title: Treatments for Fathers With Attention Deficit/Hyperactivity Disorder (ADHD) and Their At-Risk Children (Fathers Too)
Brief Title: Treatments for Fathers With ADHD and Their At-Risk Children (Fathers Too)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Mark Stein, PI, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fathers Too
Record Dates: First submitted 2016-01-20; First posted 2016-02-05 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Attention Deficit/Hyperactivity Disorder (ADHD)
Keywords: ADHD; ADD; Attention Deficit/Hyperactivity Disorder; Attention; Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm | interventions — Lisdexamfetamine Dimesylate; Methylphenidate; 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medication Arm (Active Comparator): Vyvanse Arm: 3-week open-label titration beginning at 20 mg Vyvanse (a class II drug), and be increased weekly during the titration period until an optimal response is obtained and then continue for 5 weeks. Optimal response is defined as a clinician Clinical Global Impression-Improvement score (CGI-I) ≤ 2 with minimal associated adverse events. Fathers will remain on optimal dose through the course of the study. In cases of poor tolerability or loss of efficacy the dose can be changed. If an optimal response is not achieved a trial with a long acting methylphenidate will be initiated based upon the Texas algorithm for stimulant medication. The study physician will be available by phone 24 hours/day; participants will be instructed to call with any safety concerns.
  Interventions: Drug: Vyvanse; Drug: Methylphenidate
- Behavioral Parent Training Arm (Active Comparator): Behavioral Parent Training (BPT) Arm: Fathers in the BPT group will receive weekly parent training sessions based on the Barkley manual, "Defiant Children, Third Edition". The child participants will also come to several sessions at the clinician's and supervisor's discretion.
  Interventions: Behavioral: Behavioral Parent Training

INTERVENTIONS:
Drug: Vyvanse — Half of the participants (fathers) will be randomized to receive Vyvanse.
  Other Names: lisdexamfetamine dimesylate
  Arms: Medication Arm
Behavioral: Behavioral Parent Training — Half of the fathers will receive behavioral parent training.
  Other Names: BPT
  Arms: Behavioral Parent Training Arm
Drug: Methylphenidate — If Vyvanse is not well tolerated, methylphenidate can be prescribed.
  Other Names: MPH
  Arms: Medication Arm

SUMMARY:
In contrast to mothers with Attention Deficit/Hyperactivity Disorder (ADHD), the impact of paternal ADHD in families and children with ADHD symptoms has not been studied, despite the prevalence of ADHD in males. Thus, the investigators do not know the feasibility, impact on treatment on the family and child, and effects of treating fathers relative to mothers with ADHD. Paternal ADHD is associated with negative parenting and child conduct problems.

The investigators hypothesize that successfully treating parental ADHD in fathers will have a beneficial effects on the family that will extend to the child. Specifically, the investigators believe that stimulant medication ((Lisdexamfetamine (LDX) or a different ADHD medication if poor response to LDX) with fathers will reduce father's ADHD symptoms and improve parenting. Effects of stimulant treatment of fathers will be compared to Behavioral Parent Training (BPT) on parenting, and paternal and child outcomes in fathers with ADHD who have children between the ages of 3 -8.

As in the investigator's previous work, the investigators will bank paternal and child DNA and RNA for later examination of pharmacogenetic and epigenetic effects (i.e. RNA) of stimulant response.

DETAILED DESCRIPTION:
The overarching goal of this research program is to construct and evaluate paternal and familial interventions to improve the trajectory of ADHD outcomes in at-risk young children with ADHD symptoms who have not yet been treated with stimulant medications. These children are at risk for ADHD by virtue of paternal ADHD and maladaptive parenting. Our primary outcome measure for the child will be whether child ADHD symptoms on the Conners Parent and Teacher Rating Scales decreased at the completion of the study. The primary outcomes for the fathers will be the Conners Adult ADHD Rating Scale-Self Report and Other Report (CAARS), the clinician completed Clinical Global Impressions-Severity (CGI-S) and the Barkley Functional Impairment rating Scale (BFIS). Secondary outcomes include the Family Routines Questionnaire (FRI), the Alabama Parent Questionnaire (APQ) and the Dyadic Parent-Child Interaction Coding System (DPICS).

Specific Aim 1: To develop screening and recruitment strategies for identifying fathers with ADHD who have young children at risk for ADHD.

Specific Aim 2: To assess the comparative efficacy of treating fathers with LDX (or a different ADHD medication if poor response to LDX) and functional impairment after 8 weeks of treatment.

Hypothesis 1a: LDX will be associated with a greater reduction in paternal ADHD symptoms (CAARS, CAARS-Other Informant) and impairment (CGI-S) than families treated with BPT.

Hypothesis 1 b: BPT will be associated with greater improvement on measures of parenting (e.g. APQ, DPICS) and family functioning (DAS, BFIS) than LDX.

To the investigator's knowledge, this 2.5 year study will be the very first to examine the benefit of identifying and treating fathers with ADHD prior to treating the at-risk child. In addition, to the investigator's knowledge, this is the first study to directly compare the impact of BPT vs. LDX on both father and child outcomes. Thus, the investigator's propose a novel treatment strategy for a not uncommon but difficult to treat patient population: young children who are at risk for ADHD by virtue of their early-onset behavior problems and environmental factors such a poor parenting.

ELIGIBILITY:
Fathers Inclusion Criteria:

* Sign informed consent
* Be between 21-55 years old (inclusive) at the screening visit
* English-speaking
* At screening (after washout, if required) meet full DSM-IV criteria for ADHD, any subtype
* Current CGI-S-ADHD rating ≥ 4 and < 7.
* Findings on physical exam (PE), laboratory studies, vital signs, and electrocardiogram (ECG) judged to be normal for age with no contraindications for MPH treatment.
* Pulse and blood pressure (BP) within 95% of age and gender mean
* Commit to the entire visit schedule for the study.
* Able to complete all study assessments.
* Fathers with comorbid mood/anxiety disorders which are effectively treated with antidepressants or anti-anxiety agents will be eligible for participation, provided this medication has not changed within 30 days, is well tolerated, and that current mood symptoms are not severe or associated with active suicidal ideation.

Father Exclusion Criteria:

* History of allergic reactions or severe negative response to study medications
* Active alcohol/substance abuse in the past 3 months or a positive urinary toxic screen on initial evaluation that is not explained by a time-limited medical circumstance.
* Current bipolar illness, schizophrenia, psychoses, or significant suicidal risk
* History of chronic or acute medical disorder for which stimulant therapy would be contraindicated (e.g., glaucoma, hypertension).
* Currently, (or within the past 30 days) receiving stimulant medication for ADHD.
* Father should not seek parent-based interventions during the course of the study, Weeks 1 - 8.

Child Inclusion Criteria:

* Sign assent if older than six.
* Be between the ages of 3-8.
* Symptoms of ADHD (Conners Hyperactivity Index or Attention > 60).
* English speaking.
* No prior treatment with effective doses of stimulants.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
CGI -S - ADHD rating scale (Father) | Change from Screening at 8 weeks.
  Clinical Global Impression - Severity .
Conners Adult ADHD Rating Scale - Self Report (Father) | Change from Screening at 8 weeks.
  This is a 93-item, reliable and valid measure assessing the core features of DSM-IV ADHD, while adding content unique to the adult expression of ADHD
Conners Other Report (about Father) | Change from Screening at 8 weeks
  Completed by collateral informant. The Conners Other Report is a reliable and valid measure assessing the core features of DSM-IV ADHD, while adding content unique to the adult expression of ADHD
Barkley Functional Impairment Rating Scale (Father) | Change from Screening at 8 weeks.
  The BFIS is a promising measure of impairment associated with adult ADHD, with adequate reliability, criterion validity with other measures of impairment, and normative data for adults. Normative data and reliable change index will allow for assessing functioning in domains relevant to the current proposal (i.e. Home-family, Daily Responsibilities, Child Rearing) as Well as Mean Impairment Score are sensitive to treatment effects.
Conners Parent (completed by parent about child) | Change form Screening at 8 weeks.
  Conners Parent Rating Scale that results in factor scores for Oppositional Behavior, Cognitive Problems, and Hyperactivity. There is extensive normative data and evidence of reliability, validity, and clinical utility (Hart, 1999). This will be the primary measure specifically for ADHD and externalizing symptoms.
Conners Teacher Rating Scale (completed by teacher about child) | Change from Screening at 8 weeks.
  Conners Teacher Rating Scale that results in factor scores for Oppositional Behavior, Cognitive Problems, and Hyperactivity. There is extensive normative data and evidence of reliability, validity, and clinical utility (Hart, 1999). This will be the primary measure specifically for ADHD and externalizing symptoms.

SECONDARY OUTCOMES:
Barkley Functional Impairment Rating Scale (BFIS) - Other | Change from Baseline at 8 Weeks.
  Completed by collateral informant. The BFIS is a promising measure of impairment associated with adult ADHD, with adequate reliability, criterion validity with other measures of impairment, and normative data for adults. Normative data and reliable change index will allow for assessing functioning in domains relevant to the current proposal (i.e. Home-family, Daily Responsibilities, Child Rearing) as Well as Mean Impairment Score are sensitive to treatment effects.
Family Routines Inventory (FRI) | Change from Baseline at 8 Weeks.
  The FRI is a 26-item parent-report measure that assesses the frequency with which families engage in a broad range of routines.
Alabama Parenting Questionnaire (APQ) | Change from Baseline at 8 Weeks.
  is a 42-item measure on which parents are asked to indicate the frequency with which they implement the following parenting practices: Corporal Punishment, Inconsistent Discipline, Poor Monitoring/Supervision, Involvement, and Positive Parenting.
Dyadic Parent-Child Interactions (DPICS) | Change from Baseline at 8 Weeks.
  Parents and children will engage in 3 tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Stein, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
participants will receive an study report at the end of the study.

REFERENCES:
- [Derived] Boesen K, Paludan-Muller AS, Gotzsche PC, Jorgensen KJ. Extended-release methylphenidate for attention deficit hyperactivity disorder (ADHD) in adults. Cochrane Database Syst Rev. 2022 Feb 24;2(2):CD012857. doi: 10.1002/14651858.CD012857.pub2. PMID 35201607